CLINICAL TRIAL: NCT06775613
Title: Solving Challenging Diagnoses Through Ultra-long Read Sequencing
Acronym: SCHeDULeRS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SCHeDULeRS; Horizon 2020 (Other Grant/Funding Number: European Commission)
Record Dates: First submitted 2024-11-28; First posted 2025-01-15 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-01

CONDITIONS: Variant Nucleotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Target (Experimental): Sequencing in samples with alterations in the PKD1 or CYP21A2 genes or with deletions identified by aCGH, LRS will be limited to the genes/loci of of interest.
  Interventions: Genetic: Long-read sequencing
- Genomics (Experimental): The entire genome will be analysed in samples with duplications in order to precisely identify the genomic regions in which the duplicated portions have inserted
  Interventions: Genetic: Long-read sequencing

INTERVENTIONS:
Genetic: Long-read sequencing — The technology performed belongs to third-generation sequencing strategies and is capable of analysing very long DNA and RNA fragments.

SUMMARY:
If the study is able to demonstrate that the LRS concretely overcomes the technical limitations of diagnostic methods routinely used in laboratories, its clinical application may make possible a more accurate analysis of repeated genomic regions and offer greater sensitivity for identifying SVs (Structural Variants)

DETAILED DESCRIPTION:
The diagnostic performance of LRS, by applying Oxford Nanopore Technology (ONT), will be evaluated through a real-time targeted approach and generation of ultra-long reads, to the identification of pathogenetic variants in genetic disorders with a currently challenging diagnosis due to the presence of pseudogenes (1) and to the precise mapping of SV breakpoints identified by aCGH for the definition of their clinical significance (2).

1. Patients with an established molecular diagnosis will be collected for each of the following disorders: 10 with autosomal dominant polycystic kidney disease (ADPKD) and 10 with CYP21 deficiency. Cases with ambiguous results to test possible ONT improvements in terms of time to results and precise molecular characterization will be included. The entire range of mutations affecting each causative gene (PKD1 and CYP21A2, respectively), which globally cover all the possible types of alterations (missense, nonsense, indels, exonic and gene deletions) will be included.
2. Collection of other 10 patients carrying copy number variants (CNVs) with aCGH-defined breakpoints mapping close to disease-genes possibly responsible for the observed clinical picture.

The main aim of this proposal is to evaluate ONT efficacy in resolving diagnostic challenges faced in the clinical genomics routine, in situations when a precise molecular diagnosis is often impossible or difficult and extremely time-consuming with current genetic tests. Sanger sequencing, NGS panels and MLPA are routinely used to identify pathogenic variants and CNVs responsible for many monogenic disorders and for the analysis through aCGH patients with isolated or syndromic intellectual disability without a specific clinical suspect. These analyses are long, technically laborious and often not individually conclusive because technical limitations may lead to ambiguous results and prevent definite diagnosis. The intent is to demonstrate that ONT, through a real-time targeted approach to increase coverage in clinically relevant regions during sequencing, outperforms current diagnostic tools in terms of rapidity and sensitivity, considerably improving the efficiency of the diagnostic process. The success of the proposed target ONT approach will provide the proof of principle to implement this strategy for the diagnosis of a wider spectrum of disorders already studied in our laboratory

ELIGIBILITY:
Inclusion criteria

* Patients with pathogenic alterations in the PKD1 gene, aged between 30 and 70 years
* Patients with pathogenic alterations in the CYP21A2 gene or with a not clearly defined genotype, aged between one month and 50 years
* Patients carrying potentially pathogenic CNVs (e.g. new onset and/or in proximity of disease-associated genes), aged between one month up to 70 years
* Availability of a suitable blood sample at the IRCCS Medical Genetics Unit AOUBO
* Acquisition of informed consent.

Exclusion criteria

- None

Ages: 28 Days to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Genetic anomalies | 24 months
  To determine the sensitivity of the LRS in detectiong genetic variants in hard-to-analyze genomic regions and to enables precise mapping of unbalanced genomic alterations identified by routine diagnostic techniques.

SECONDARY OUTCOMES:
Mapping the breaking points of CNVs | 24 months
  To verify whether the new sequencing technology impacts the analysis and reporting times.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Magini, Biologist, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No